CLINICAL TRIAL: NCT06519045
Title: Pharmacokinetic Profiles of Codeine and Metabolites in Fingerprint Sweat, Oral Fluid, Blood and Urine Following Controlled, Oral Administration of Codeine Phosphate Tablets to 40 Healthy Adults
Brief Title: PK of Codeine and Metabolites in Human Fingerprint Sweat, Oral Fluid, Blood and Urine
Status: Active, not recruiting | Type: Observational
Sponsor: Intelligent Bio Solutions Inc. (Industry)
Collaborators: Cliantha Research (Other)
Responsible Party: Sponsor
Other Study IDs: IBS-2024-01
Record Dates: First submitted 2024-06-17; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Pharmacokinetics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fingerprint sweat, oral fluid, whole blood, and urine specimens will be collected. No DNA analysis will take place.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- 1: Dosed with 3x60mg codeine
  Interventions: Device: Intelligent Fingerprinting Drug Screening System

INTERVENTIONS:
Device: Intelligent Fingerprinting Drug Screening System — The Intelligent Fingerprinting Drug Screening System utilizes a single-use, rapid, non-invasive fingerprint sweat drug screening test intended for use with the Intelligent Fingerprinting DSR-Plus fluorescence reader. The Intelligent FingerprintingTM Fingerprint Collection Kit for Laboratory Analysis (i.e. confirmation test) provides a quantitative analytical result via laboratory-based liquid chromatography/tandem mass spectrometry (LC-MS/MS). It is used to collect and measure drug mass in the full set of 10 fingerprints.

SUMMARY:
This study will compare positive and negative test results obtained from fingerprint sweat using the Intelligent Fingerprinting Drug Screening Cartridge, versus opiates in sweat collected via the Fingerprint Collection Kit for Laboratory Analysis, versus blood, oral fluid and urine sample concentrations of opiates identified within codeine phosphate dosed healthy males and non-pregnant females.

ELIGIBILITY:
Inclusion Criteria:

1. Informed of the nature of the study, agreed to, and able to read, review, and sign the informed consent document prior to dosing.
2. Completed the IRB-approved screening process within 28 days prior to dosing.
3. Healthy male and non-pregnant female subjects between ages 18 and 55, inclusive, at the time of dosing.
4. Body mass index (BMI) between 18 kg/m2 to 32 kg/m2, inclusive, and weigh at least 60 kg.
5. Judged by the Investigator and/or designee to be in good health as documented by the medical history, physical examination, clinical laboratory assessments, and by general observations.
6. Subjects with glomerular filtration rate (GFR) of greater than or equal to 60.
7. Females of childbearing potential must be willing to practice an acceptable form of contraception, and have a negative serum pregnancy test at screening and a negative urine pregnancy test on admission to the treatment phase of the study.
8. Males must agree to practice an acceptable form of contraception.

Exclusion Criteria:

1. More than three digits absent from the hands due to congenital or accidental cause(s).
2. Reports receiving any investigational drug/product within 30 days prior to dosing.
3. Reports any personal history of substance abuse (including drug/alcohol abuse or addiction) or mental illness (e.g. major depression) within one year prior to screening visit.
4. Reports any presence or history of a clinically significant disorder involving the cardiovascular, respiratory, renal, urologic, gastrointestinal, hepatic, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease as determined by the Investigator.
5. Presence of any clinically significant results from laboratory tests, vital signs assessments, and electrocardiograms, as judged by the Investigator.
6. Demonstrates a reactive screen for hepatitis B surface antigen, hepatitis C antibody, or HIV antibody.
7. Reports a clinically significant illness during the 28 days prior to dosing (as determined by the Investigator).
8. Reports a history of allergic response(s) to Naltrexone or other opiates/related drugs.
9. Reports hypersensitivity to bisulfites.
10. Reports history of respiratory depression (e.g., sleep apnea).
11. Current severe hypotension (i.e., systolic blood pressure <90 mmHg).
12. Reports current presence of acute bronchial asthma/ upper airway obstruction.
13. If subject reports a history of clinically significant allergies, including food or drug allergies, as judged by the Investigator.
14. Reports history/current condition of adrenal insufficiency.
15. Reports history/current condition of renal disease.
16. Demonstrates a positive drug screen for cotinine or history of smoking within previous six months.
17. Report history/current condition of seizures, increased intracranial pressure, brain tumor, head injuries or impaired consciousness.
18. Reports a blood donation totaling between 101 mL to 499 mL of blood within 30 days prior to dosing or subject who has donated more than 499 mL of blood within 56 days prior to dosing. All subjects will be advised not to donate blood for 30 days after completing the study.
19. Reports donating plasma (e.g., plasmapheresis) within 14 days prior to dosing. All subjects will be advised not to donate plasma for 30 days after completing the study.
20. Demonstrates, in the opinion of study staff, veins unsuitable for repeated venipuncture (e.g., veins difficult to locate, access, or puncture; veins with a tendency to rupture during or after puncture).
21. Reports known or suspected gastrointestinal obstruction including, paralytic ileus.
22. Reports difficulty fasting or consuming standardized meals.
23. Demonstrates a positive pregnancy screen (females only).
24. If, in the opinion of the Investigator, the subject is not suitable for the study.

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: Subjects will be selected from non-institutionalized subjects consisting of members of the community at large.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) of codeine and codeine-6-glucuronide in fingerprint sweat, oral fluid, plasma, and urine | From -1 hr to 24 hrs relative to codeine sulfate dose
  Peak concentration in each of fingerprint sweat, oral fluid, plasma, and urine, as calculated from LC-MS/MS analysis of specimens
Time to reach maximum concentration (Tmax) of codeine and codeine-6-glucuronide in fingerprint sweat, oral fluid, plasma, and urine | From -1 hr to 24 hrs relative to codeine sulfate dose
  Time after drug administration at which peak plasma concentration occurs in each of fingerprint sweat, oral fluid, plasma, and urine, as calculated from LC-MS/MS analysis of specimens
Area under the curve (AUC) of codeine in fingerprint sweat, oral fluid, plasma, and urine | From -1 hr to 24 hrs relative to codeine sulfate dose
  Efficiency of physiological processes that characterize the drug elimination in each of fingerprint sweat, oral fluid, plasma, and urine, as calculated from LC-MS/MS analysis of codeine and codeine-6-glucuronide in specimens
Terminal half-life (T1/2) of codeine in fingerprint sweat, oral fluid, plasma, and urine | From -1 hr to 24 hrs relative to codeine sulfate dose
  The period of time that it takes for the concentration of codeine and codeine-6-glucuronide to decrease by 50% in each of fingerprint sweat, oral fluid, plasma, and urine, as calculated from LC-MS/MS analysis of codeine and codeine-6-glucuronide in specimens
Clearance of codeine in fingerprint sweat, oral fluid, plasma, and urine | From -1 hr to 24 hrs relative to codeine sulfate dose
  Amount of codeine eliminated per unit of time/ drug concentration in each of fingerprint sweat, oral fluid, plasma, and urine, as calculated from LC-MS/MS analysis of codeine and codeine-6-glucuronide in specimens

SECONDARY OUTCOMES:
Sensitivity of fingerprint sweat screening system for codeine | From -1 hr to 24 hrs relative to codeine sulfate dose
  Comparison of results of fingerprint sweat screening system to LC-MS/MS analysis of fingerprint sweat specimens for codeine

CONTACTS AND LOCATIONS:
Overall Officials: Philip Mathew, MD, Principal Investigator — Cliantha Research
Locations (1):
- Cliantha Research, Mississauga, Ontario, Canada